CLINICAL TRIAL: NCT05627219
Title: Peer Genetic Coaches for Enhancing Genetic Testing Awareness, Navigation, and Delivery Among African American Men With Metastatic Prostate Cancer, The EXPAND Network
Brief Title: Extending Prostate Genetic Awareness, Navigation, and Delivery: The EXPAND Network
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 22C.423; JT 22046 (Other: JeffTrial Number)
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Prostate Carcinoma; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Educational Status; Early Intervention, Educational; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Supportive care (training, education, discussion): AIM 1: Peer genetic coaches undergo training and education on study.
  AIM 2: Patients receive an educational booklet and attend a discussion with a peer genetic coach on study.
  Interventions: Behavioral: Training and Education; Other: Educational Intervention; Procedure: Discussion

INTERVENTIONS:
Behavioral: Training and Education — Undergo training and education
Other: Educational Intervention — Receive educational booklet
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention; Educational
Procedure: Discussion — Attend discussion with peer genetic coach
  Other Names: Discuss

SUMMARY:
This trial evaluates whether a network of peer genetic coaches is useful for addressing disparities in genetic testing and screening among African American men with prostate cancer that has spread from where it first started (primary site) to other places in the body (metastatic). While genetic testing has become central to prostate cancer care, African American men are less likely seek testing due to lack of awareness, cultural beliefs, financial limitations, fear of discrimination, and mistrust in the healthcare system. A network of peer genetic coaches may help address barriers, beliefs, and needs of African American men in the community and provide navigation to increase engagement in genetic testing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify and train 6 African American (AA) men as peer genetic coaches (PGCs) for the Extending Prostate Genetic Awareness, Navigation, and Delivery (EXPAND) Network. (Train peer genetic coaches) II. Conduct a feasibility study of peer genetic coaching. (Provide individual coaching)

SECONDARY OBJECTIVE:

I. Patient-related outcomes will include change in decisional conflict for genetic counseling, acceptability/attitude toward genetic counseling and testing, and change of genetics knowledge.

OUTLINE:

AIM 1: Peer genetic coaches undergo training and education on study.

AIM 2: Patients receive an educational booklet and attend a discussion with a peer genetic coach on study.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Are 18 years old or older
* AIM 1: Are able to read and speak English comfortably
* AIM 1: Men who have experience with both prostate cancer (PCA) and genetic counseling and testing will be a priority for training, as well as men who have considerable peer education or navigation experience
* AIM 2: Are 18 years old or older
* AIM 2: Are African American
* AIM 2: Are able to read and speak English comfortably
* AIM 2: Men who meet any one of the following criteria: (1) metastatic prostate cancer; (2) prostate cancer with high-risk features (T3 or higher, Gleason 8 or higher, node positive disease); (3) with or without a diagnosis of prostate cancer with strong family history (2 or more first-degree or second-degree relatives) with prostate cancer (particularly metastatic prostate cancer or died from prostate cancer), breast cancer, ovarian cancer, pancreatic cancer, colorectal cancer, uterine cancer, renal cancer, urothelial cancer, or upper bowel cancer

Exclusion Criteria:

* Patients that do not meet the inclusion criteria
* Children under the age of 18
* Anyone who has trouble understanding the consent or with significant anxiety detected during the consent process

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Men who have experience with both prostate cancer (PCA) and genetic counseling and testing, as well as peer education or navigation experience. African American men with a history of prostate cancer or with a strong family history of prostate cancer, breast cancer, ovarian cancer, pancreatic cancer, colorectal cancer, uterine cancer, renal cancer, urothelial cancer, or upper bowel cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Number of inquiries to the central number (feasibility) | Up to 1 year
Percent of callers screened and eligible to participate (feasibility) | Up to 1 year
Percent of eligible callers who enroll in the study (feasibility) | Up to 1 year
Percent who complete the endpoint assessment (feasibility) | Up to 1 year
Number and percent of men making genetic counseling appointments | Up to 1 year

SECONDARY OUTCOMES:
Change in decisional conflict for genetic counseling | Baseline up to 1 year
  Reported with mean and standard deviation.
Change in acceptability/attitude toward genetic counseling and testing | Baseline up to 1 year
  Reported with mean and standard deviation.
Change of genetics knowledge | Baseline up to 1 year
  Reported with mean and standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Amy Leader, DrPh, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No